CLINICAL TRIAL: NCT02228382
Title: A PHASE 4 SAFETY AND EFFICACY STUDY OF BOSUTINIB (BOSULIF (REGISTERED)) IN PATIENTS WITH PHILADELPHIA CHROMOSOME POSITIVE CHRONIC MYELOID LEUKEMIA PREVIOUSLY TREATED WITH ONE OR MORE TYROSINE KINASE INHIBITORS
Brief Title: Safety And Efficacy Study Of Bosutinib In Patients With Philadelphia Chromosome Positive Chronic Myeloid Leukemia Previously Treated With One Or More Tyrosine Kinase Inhibitors
Status: Terminated | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer (Industry)
Collaborators: Developmental Therapeutics Consortium (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Masking: None | Purpose: Treatment
Other Study IDs: B1871039; 2013-003250-25 (EudraCT Number); BYOND (Other: Alias Study Number)
Record Dates: First submitted 2014-08-27; First posted 2014-08-29 (Estimated); Results first posted 2021-12-30 (Actual); Last update posted 2021-12-30 (Actual); Status verified 2021-12

CONDITIONS: Previously Treated PH + CML
Keywords: Bosutinib; Chronic Myeloid Leukemia; CML; Leukemia; Myelogenous; Chronic; BC-ABL Positive
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Leukemia; Bronchiolitis Obliterans Syndrome | interventions — bosutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Bosutinib (Experimental)
  Interventions: Drug: Bosutinib

INTERVENTIONS:
Drug: Bosutinib — 100 mg and 500 mg tablets, once daily dosage up to 4 years duration
  Other Names: BOSULIF

SUMMARY:
The purpose of this study is to fulfill the post-authorization commitment made by Pfizer to the European Medicines Agency in providing additional safety and efficacy data in approximately 150 Philadelphia Chromosome Positive Chronic Myeloid Leukemia patients with high unmet medical need, including 75 Chronic Phase, Accelerated Phase or Blast Phase patients in the fourth or later line treatment setting (i.e., after treatment with at least 3 other Tyrosine Kinase Inhibitors).

ELIGIBILITY:
Inclusion Criteria:

* Confirmed Philadelphia Chromosome positive Chronic Myeloid Leukemia or Confirmed BCR-ABL1 (Abelson-break point cluster) Positive if Philadelphia Chromosome negative Chronic Myeloid Leukemia (from initial diagnosis).
* Prior treatment with 1 or more tyrosine kinase inhibitor drugs (imatinib, dasatinib and/or nilotinib) for Philadelphia Chromosome positive Chronic Myeloid Leukemia (CML).
* Any Chronic Myeloid Leukemia disease phase, as long as the patient is unable to receive treatment with imatinib, dasatinib and/or nilotinib for any reason.

Exclusion Criteria:

* Participation in any other clinical studies involving investigational drug(s) within 14 days or within 3 half-lives of drug levels in blood (whichever is longer) prior to the first dose of bosutinib.
* Prior treatment with bosutinib.
* Prior treatment with ponatinib.
* Known T315I or V299L mutation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 163 (Actual)
Dates: Start 2014-11-07 (Actual); Primary Completion 2020-10-13 (Actual); Study Completion 2020-10-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (48):
- United States (13):
  - Keck Hospital of USC, Los Angeles, California
  - LAC+USC Medical Center, Los Angeles, California
  - USC/Norris Comprehensive Cancer Center, Los Angeles, California
  - Sylvester Deerfield Beach, Deerfield Beach, Florida
  - University of Miami Hospital & Clinics, Miami, Florida
  - Indiana Blood and Marrow Transplantation-Clinic, Indianapolis, Indiana
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Siteman Cancer Center - West County, Creve Coeur, Missouri
  - Barnes-Jewish Hospital, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Siteman Cancer Center - South County, St Louis, Missouri
  - Weill Cornell Medical College - New York-Presbyterian Hospital, New York, New York
  - Seattle Cancer Care Alliance, Seattle, Washington
- Austria (2):
  - Medizinische Universitaet Innsbruck, Innsbruck
  - Ordensklinikum Linz Gmbh Barmherzige Schwestern, Linz
- France (6):
  - Institut Bergonie, Bordeaux
  - Centre Hospitalier de Versailles (CHV)-Hopital Andre Mignot Service d'Hematologie Clinique- Oncology, Le Chesnay
  - Centre Regional De Lutte Contre Le Cancer, Marseille
  - Hopital Archet I, Nice
  - Institut Universitaire du Cancer Toulouse - Oncopole, Toulouse
  - CHU Brabois, Vandœuvre-lès-Nancy
- Germany (6):
  - RWTH Uniklinik Aachen Klinik fur Onkologie, Hamatologie und Stammzelltransplantation, Aachen
  - Charite - Universitaetsmedizin Berlin - Campus Virchow-Klinikum (CVK), Berlin
  - Universitaetsklinikum Koeln (AoeR), Cologne
  - Universitaetsklinikum Hamburg-Eppendorf, Hamburg
  - Klinik fur Innere Medizin II, Jena
  - III. Medizinische Klinik Universitaetsmedizin Mannheim, Mannheim
- Italy (8):
  - AOU Policlinico Consorziale di Bari - UO Ematologia con Trapianto, Bari, BA
  - A.O.U. Policlinico S. Orsola-Malpighi, Bologna, BO
  - Azienda Socio Sanitaria Territoriale - ASST Monza, Monza, MB
  - Ospedale S. Eugenio - UOC Ematologia, Rome, RM
  - AOU San Luigi Gonzaga SCDU Medicina Interna II ad indirizzo Ematologico, Orbassano, TO
  - AOU Policlinico Vittorio Emanuele-P.O.G. Rodolico, Catania
  - SOD Ematologia, Florence
  - A.O. Ospedale Niguarda Ca Granda - SC Ematologia, Milan
- Norway (2):
  - Haukeland Universitetssjukehus, Bergen
  - St Olav Hospital, Trondheim
- Spain (9):
  - Hospital Universitario Quiron Madrid, Pozuelo de Alarcón, Madrid
  - Hospital Universitari Vall d' Hebron, Barcelona
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Clinic De Barcelona, Barcelona
  - Hospital Universitario de La Princesa, Madrid
  - Hospital Universitario Ramon y Cajal, Madrid
  - Hospital Clinico Universitario de Salamanca, Salamanca
  - Hospital Universitari i Politecnic La Fe de Valencia, Valencia
  - Hospital de dia Quiron Zaragoza, Zaragoza
- Sweden (2):
  - Hematologiskt centrum, Stockholm
  - Akademiska Sjukhuset, Uppsala

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Gambacorti-Passerini C, Brummendorf TH, Abruzzese E, Kelly KR, Oehler VG, Garcia-Gutierrez V, Hjorth-Hansen H, Ernst T, Leip E, Purcell S, Luscan G, Viqueira A, Giles FJ, Hochhaus A. Efficacy and safety of bosutinib in previously treated patients with chronic myeloid leukemia: final results from the BYOND trial. Leukemia. 2024 Oct;38(10):2162-2170. doi: 10.1038/s41375-024-02372-x. Epub 2024 Aug 20. PMID 39164407
- [Derived] Smith BD, Brummendorf TH, Roboz GJ, Gambacorti-Passerini C, Charbonnier A, Viqueira A, Leip E, Purcell S, Goldman EH, Giles F, Ernst T, Hochhaus A, Rosti G. Efficacy and safety of bosutinib in patients treated with prior imatinib and/or dasatinib and/or nilotinib: Subgroup analyses from the phase 4 BYOND study. Leuk Res. 2024 Apr;139:107481. doi: 10.1016/j.leukres.2024.107481. Epub 2024 Mar 11. PMID 38484432
- [Derived] Rosti G, Brummendorf TH, Gjertsen BT, Giraldo-Castellano P, Castagnetti F, Gambacorti-Passerini C, Ernst T, Zhao H, Kuttschreuter L, Purcell S, Giles FJ, Hochhaus A. Impact of age and comorbidities on the efficacy and tolerability of bosutinib in previously treated patients with chronic myeloid leukemia: results from the phase 4 BYOND study. Leukemia. 2024 Jan;38(1):126-135. doi: 10.1038/s41375-023-02080-y. Epub 2023 Nov 25. PMID 38007586
- [Derived] Takahashi N, Cortes JE, Sakaida E, Ishizawa K, Ono T, Doki N, Matsumura I, Garcia-Gutierrez V, Rosti G, Ono C, Ohkura M, Tanetsugu Y, Viqueira A, Brummendorf TH. Safety profile of bosutinib in Japanese versus non-Japanese patients with chronic myeloid leukemia: a pooled analysis. Int J Hematol. 2022 Jun;115(6):838-851. doi: 10.1007/s12185-022-03314-y. Epub 2022 Mar 2. PMID 35235189
- [Derived] Hochhaus A, Gambacorti-Passerini C, Abboud C, Gjertsen BT, Brummendorf TH, Smith BD, Ernst T, Giraldo-Castellano P, Olsson-Stromberg U, Saussele S, Bardy-Bouxin N, Viqueira A, Leip E, Russell-Smith TA, Leone J, Rosti G, Watts J, Giles FJ; BYOND Study Investigators. Bosutinib for pretreated patients with chronic phase chronic myeloid leukemia: primary results of the phase 4 BYOND study. Leukemia. 2020 Aug;34(8):2125-2137. doi: 10.1038/s41375-020-0915-9. Epub 2020 Jun 22. PMID 32572189
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B1871039&StudyName=Safety%20And%20Efficacy%20Study%20Of%20Bosutinib%20In%20Patients%20With%20Philadelphia%20Chromosome%20Positive%20Chronic%20Myeloid%20Leukemia%20Previously%20Treated%20With%20

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants with chronic phase (CP), accelerated phase (AP), or blast phase (BP) philadelphia chromosome positive (Ph+) chronic myelogenous leukemia (CML), or breakpoint cluster region-abelson kinase (BCR-ABL1) positive and Philadelphia chromosome negative (Ph-), who failed prior treatment with commercially available tyrosine kinase inhibitors (TKIs) due to drug resistance or intolerance, or were otherwise contraindicated for treatment with commercially available TKIs were enrolled.
Pre-assignment Details: A total of 177 participants signed the ICF, 14 participants were screen failure and 163 were enrolled into the study and assigned to study treatment. Reporting arms were based on line of therapy (CP2L, CP3L, CP4L) and disease phase (CP and AP). Data collection and planned analysis on BP participants was not performed because no participants with BP were enrolled in the study.
Groups:
- Bosutinib: Chronic Phase 2nd Line Chronic Myelogenous Leukemia: Participants with philadelphia chromosome positive chronic phase 2nd line chronic myelogenous leukemia resistant or intolerant to imatinib, dasatinib, or nilotinib received bosutinib 500 milligram (mg), orally once daily until disease progression, unacceptable toxicity, withdrawal of consent, death or discontinuation of study (up to maximum of 4 years). Participants who discontinued bosutinib prior to completing at least 4 years of therapy were followed for survival until they completed at least 4 years of follow-up from the time of first dose.
- Bosutinib: Chronic Phase 3rd Line Chronic Myelogenous Leukemia: Participants with philadelphia chromosome positive chronic Phase 3rd line chronic myelogenous leukemia resistant or intolerant to imatinib and/or dasatinib and/or nilotinib received bosutinib 500 mg, orally once daily until disease progression, unacceptable toxicity, withdrawal of consent, death or discontinuation of study (up to maximum of 4 years). Participants who discontinued bosutinib prior to completing at least 4 years of therapy were followed for survival until they completed at least 4 years of follow-up from the time of first dose.
- Bosutinib: Chronic Phase 4th Line Chronic Myelogenous Leukemia: Participants with philadelphia chromosome positive chronic phase 4th line chronic myelogenous leukemia resistant or intolerant to imatinib and dasatinib and nilotinib received bosutinib 500 mg, orally once daily until disease progression, unacceptable toxicity, withdrawal of consent, death or discontinuation of study (up to maximum of 4 years). Participants who discontinued bosutinib prior to completing at least 4 years of therapy were followed for survival until they completed at least 4 years of follow-up from the time of first dose.
- Bosutinib: Accelerated Phase Chronic Myelogenous Leukemia: Participants with philadelphia chromosome positive accelerated phase chronic myelogenous leukemia resistant or intolerant to at least one tyrosine kinase inhibitor among imatinib, dasatinib, or nilotinib received bosutinib 500 mg, orally once daily until disease progression, unacceptable toxicity, withdrawal of consent, death or discontinuation of study (up to maximum of 4 years). Participants who discontinued bosutinib prior to completing at least 4 years of therapy were followed for survival until they completed at least 4 years of follow-up from the time of first dose.
- Bosutinib: Philadelphia Chromosome Negative Chronic Myelogenous Leukemia: Participants with BCR-ABL1 positive and philadelphia chromosome negative chronic myelogenous leukemia received bosutinib 500 mg, orally once daily until disease progression, unacceptable toxicity, withdrawal of consent, death or discontinuation of study (up to maximum of 4 years). Participants who discontinued bosutinib prior to completing at least 4 years of therapy were followed for survival until they completed at least 4 years of follow-up from the time of first dose.
Period: Overall Study
Arm/Group | Bosutinib: Chronic Phase 2nd Line Chronic Myelogenous Leukemia | Bosutinib: Chronic Phase 3rd Line Chronic Myelogenous Leukemia | Bosutinib: Chronic Phase 4th Line Chronic Myelogenous Leukemia | Bosutinib: Accelerated Phase Chronic Myelogenous Leukemia | Bosutinib: Philadelphia Chromosome Negative Chronic Myelogenous Leukemia
Started | 46 | 61 | 49 | 4 | 3
Completed | 36 | 43 | 28 | 2 | 1
Not Completed | 10 | 18 | 21 | 2 | 2
Not completed — Death | 5 | 7 | 5 | 0 | 2
Not completed — Participant refused further follow-up | 0 | 0 | 1 | 0 | 0
Not completed — Study terminated by sponsor | 3 | 5 | 7 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 3 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 3 | 2 | 1 | 0
Not completed — Other | 2 | 3 | 3 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety analysis set included all participants who received at least 1 dose of bosutinib
Groups:
- Bosutinib: Chronic Phase 2nd Line Chronic Myelogenous Leukemia: Participants with philadelphia chromosome positive chronic phase 2nd line chronic myelogenous leukemia.
- Bosutinib: Chronic Phase 3rd Line Chronic Myelogenous Leukemia: Participants with philadelphia chromosome positive chronic Phase 3rd line chronic myelogenous leukemia.
- Bosutinib: Chronic Phase 4th Line Chronic Myelogenous Leukemia: Participants with philadelphia chromosome positive chronic phase 4th line chronic myelogenous leukemia.
- Bosutinib: Accelerated Phase Chronic Myelogenous Leukemia: Participants with philadelphia chromosome positive accelerated phase chronic myelogenous leukemia.
- Bosutinib: Philadelphia Chromosome Negative Chronic Myelogenous Leukemia: Participants with BCR-ABL1 positive and philadelphia chromosome negative chronic myelogenous leukemia.
- Total: Total of all reporting groups
Arm/Group | Bosutinib: Chronic Phase 2nd Line Chronic Myelogenous Leukemia | Bosutinib: Chronic Phase 3rd Line Chronic Myelogenous Leukemia | Bosutinib: Chronic Phase 4th Line Chronic Myelogenous Leukemia | Bosutinib: Accelerated Phase Chronic Myelogenous Leukemia | Bosutinib: Philadelphia Chromosome Negative Chronic Myelogenous Leukemia | Total
Number analyzed (Participants) | 46 | 61 | 49 | 4 | 3 | 163
Age, Continuous [Mean (Standard Deviation); unit: Years] | 55.8 (15.4) | 61.8 (15.0) | 59.4 (15.3) | 40.8 (11.0) | 64.3 (7.1) | 58.9 (15.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 24 | 28 | 0 | 0 | 75
  Male | 23 | 37 | 21 | 4 | 3 | 88
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 0 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 2 | 1 | 1 | 0 | 0 | 4
  White | 39 | 55 | 44 | 2 | 3 | 143
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 5 | 4 | 4 | 2 | 0 | 15

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Cumulative Confirmed Major Cytogenetic Response (MCyR) in 2nd and 3rd Line Chronic Phase (CP) Participants
Description: Confirmed MCyR: confirmed (complete cytogenetic response[CCyR] or partial cytogenetic response[PCyR]) by 1 year for participants entering the study without CCyR or maintenance of confirmed CCyR for at least 1 year after treatment start with bosutinib for participants entering the study with CCyR or at least major molecular response(MMR) by 1 year and a deeper molecular response compared to baseline. Participants with baseline PCyR that did not achieve CCyR were counted as nonresponders. Initial cytogenetic (in absence of MMR) responses must have been confirmed by 2 consecutive assessments >=28 days apart. CCyR: 0% Ph+ cells from >=20 metaphases from conventional cytogenetics or <1% Ph+ cells from >= 200 cells from fluorescent in situ hybridization(FISH). PCyR: 1 to 35% Ph+ cells. MMR: <=0.1% BCR-ABL1 on the international scale (IS) with at least 10,000 ABL1 transcripts assessed by central laboratory.
Time Frame: Up to 1 year (52 weeks)
Population: Evaluable set for cytogenetic response: treated participants with valid baseline efficacy assessment (>=20 metaphases from baseline bone marrow or CCyR with >=200 cells from FISH or baseline MMR). Data for this outcome measure was not planned to be collected and analyzed for AP CML and Ph- participants and planned to be analyzed for 2nd line and 3rd line population.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Bosutinib, Chronic Phase 2nd and 3rd Line Chronic Myelogenous Leukemia: Participants with philadelphia chromosome positive chronic phase 2nd and 3rd line chronic myelogenous leukemia.
Arm/Group | Bosutinib, Chronic Phase 2nd and 3rd Line Chronic Myelogenous Leukemia
Number analyzed (Participants) | 98
percentage of participants | 76.5 [66.9 to 84.5]

2. Primary Outcome: Percentage of Participants With Cumulative Confirmed Major Cytogenetic Response (MCyR) in 4th or Later Line Chronic Phase (CP) Participants
Description: Confirmed MCyR: confirmed CCyR or PCyR by 1 year for participants entering the study without CCyR or maintenance of confirmed CCyR for at least 1 year after treatment start with bosutinib for participants entering the study with CCyR or at least MMR by 1 year and a deeper molecular response compared to baseline. Participants with baseline PCyR that did not achieve CCyR were counted as nonresponders. Initial cytogenetic (in absence of MMR) responses must have been confirmed by 2 consecutive assessments >=28 days apart. CCyR: 0% Ph+ cells from >=20 metaphases from conventional cytogenetics or <1% Ph+ cells from >= 200 cells from fluorescent in situ hybridization(FISH). PCyR: 1 to 35% Ph+ cells. MMR: <=0.1% BCR-ABL1 on the IS with at least 10,000 ABL1 transcripts assessed by central laboratory.
Time Frame: Up to 1 year (52 weeks)
Population: Evaluable set cytogenetic response: treated participants with valid baseline efficacy assessment (>= 20 metaphases from baseline bone marrow or CCyR with >=200 cells from FISH or baseline MMR). Data for this outcome measure was not planned to be collected and analyzed for AP CML and Ph-participants.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Bosutinib: Chronic Phase 4th Line Chronic Myelogenous Leukemia
Number analyzed (Participants) | 45
percentage of participants | 62.2 [46.5 to 76.2]

3. Primary Outcome: Percentage of Participants With Cumulative Confirmed Overall Hematological Response (OHR) in Accelerated Phase (AP) Chronic Myelogenous Leukemia (CML) Participants
Description: Confirmed OHR was defined as complete hematological response (CHR) or return to chronic phase (RCP) by 1 year in AP and BP participants. CHR was defined as white blood cells (WBC) <10*10^9/L, peripheral blood basophils <5%, no peripheral blood myelocytes, promyelocytes, myeloblasts in the differential, platelet count <450*10^9/L, spleen not palpable. Hematologic responses must be of >=4 weeks duration confirmed by 2 assessments >=4 weeks apart.
Time Frame: Up to 1 year (52 weeks)
Population: Evaluable set for hematological response: treated participants with a valid baseline hematologic assessment. Data for this outcome measure was not planned to be collected and analyzed for CP2L, CP3L, CP4L and Ph- CML participants.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Bosutinib: Accelerated Phase Chronic Myelogenous Leukemia
Number analyzed (Participants) | 4
percentage of participants | 75.0 [19.4 to 99.4]

4. Secondary Outcome: Percentage of Participants With Cumulative Major Cytogenetic Response (MCyR)
Description: CyR was based on prevalence of Ph+ cells. CCyR was achieved when there was 0 % Ph+ cells from >=20 metaphases from conventional bone marrow cytogenetics or <1% Ph+ cells from >=200 cells analyzed from FISH. PCyR was achieved when 1 to 35% Ph+ cells were present. MCyR was categorized as either CCyR or PCyR. Participants with MMR or better at baseline were counted as CCyR if baseline response was maintained or improved while on treatment.
Time Frame: Up to 4 years
Population: Evaluable set cytogenetic response: treated participants with valid baseline efficacy assessment (>=20 metaphases from baseline bone marrow or CCyR with >=200 cells from FISH or baseline MMR). Data for this outcome measure was not planned to be collected and analyzed for Ph- participants.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Bosutinib: Chronic Phase 2nd Line Chronic Myelogenous Leukemia | Bosutinib: Chronic Phase 3rd Line Chronic Myelogenous Leukemia | Bosutinib: Chronic Phase 4th Line Chronic Myelogenous Leukemia | Bosutinib: Accelerated Phase Chronic Myelogenous Leukemia
Number analyzed (Participants) | 43 | 55 | 45 | 4
percentage of participants | 88.4 [74.9 to 96.1] | 85.5 [73.3 to 93.5] | 77.8 [62.9 to 88.8] | 75.0 [19.4 to 99.4]

5. Secondary Outcome: Percentage of Participants With Cumulative Confirmed Overall Hematological Response (OHR) in Participants With Accelerated Phase (AP) Chronic Myelogenous Leukemia (CML)
Description: Confirmed OHR was defined as CHR or RCP in AP and BP participants. CHR was defined as WBC <10*10^9/L, peripheral blood basophils <5%, no peripheral blood myelocytes, promyelocytes, myeloblasts in the differential, platelet count <450*10^9/L, spleen not palpable. Hematologic responses must be of >=4 weeks duration confirmed by 2 assessments >=4 weeks apart.
Time Frame: Up to 4 years
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Bosutinib: Accelerated Phase Chronic Myelogenous Leukemia
Number analyzed (Participants) | 4
percentage of participants | 75.0 [19.4 to 99.4]

6. Secondary Outcome: Percentage of Participants With Cumulative Best Response
Description: Hierarchy best response: %participants with best response among molecular/cytogenetic/hematologic response. Molecular response:MR4.5/MR4/MMR defined as <=0.0032/0.01/0.1% BCR-ABL1 ratio on IS corresponding to >=4.5/4/3-log reduction from standardised baseline with at least 32,000/10,000/10,000 ABL1 assessed by central laboratory. CyR:based on prevalence of Ph+cells. CCyR: 0% Ph+cells from >=20 metaphases from conventional cytogenetics or <1%Ph+cells from >=200 cells from FISH. PCyR:1 to 35% Ph+cells. CHR:WBC <10*10^9/L, peripheral blood basophils<5%, no peripheral blood myelocytes, promyelocytes, myeloblasts in differential, platelet count<450*10^9/L, spleen not palpable.
Time Frame: Up to 4 years
Population: Evaluable set:treated participants with valid baseline molecular, cytogenetic or hematologic assessment. Data for this outcome measure (all categories including OHR) was not planned to be collected and analyzed for Ph- CML participants. Data for OHR was not planned to be collected and analyzed for CP CML participants.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Bosutinib: Chronic Phase 2nd Line Chronic Myelogenous Leukemia | Bosutinib: Chronic Phase 3rd Line Chronic Myelogenous Leukemia | Bosutinib: Chronic Phase 4th Line Chronic Myelogenous Leukemia | Bosutinib: Accelerated Phase Chronic Myelogenous Leukemia
Number analyzed (Participants) | 46 | 61 | 49 | 4
percentage of participants
  MR4.5 | 17.4 [7.8 to 31.4] | 14.8 [7.0 to 26.2] | 8.2 [2.3 to 19.6] | 25.0 [0.6 to 80.6]
  MR4 | 15.2 [6.3 to 28.9] | 11.5 [4.7 to 22.2] | 6.1 [1.3 to 16.9] | 0.0 [0.0 to 60.2]
  MMR | 8.7 [2.4 to 20.8] | 11.5 [4.7 to 22.2] | 14.3 [5.9 to 27.2] | 25.0 [0.6 to 80.6]
  CCyR | 2.2 [0.1 to 11.5] | 13.1 [5.8 to 24.2] | 14.3 [5.9 to 27.2] | 25.0 [0.6 to 80.6]
  PCyR | 2.2 [0.1 to 11.5] | 1.6 [0.0 to 8.8] | 4.1 [0.5 to 14.0] | 0.0 [0.0 to 60.2]
  CHR | 10.9 [3.6 to 23.6] | 8.2 [2.7 to 18.1] | 16.3 [7.3 to 29.7] | 0.0 [0.0 to 60.2]
  OHR: number analyzed (Participants) | 0 | 0 | 0 | 4
  OHR |  |  |  | 0.0 [0.0 to 60.2]

7. Secondary Outcome: Percentage of Participants With Major Cytogenetic Response (MCyR) at Months 3, 6, 12, 18 and 24
Description: as for outcome 4
Time Frame: Months 3, 6, 12, 18, and 24
Population: Evaluable set cytogenetic response: treated participants with valid baseline efficacy assessment (>= 20 metaphases from baseline bone marrow or CCyR with >=200 cells from FISH or baseline MMR). Data for this outcome measure was not planned to be collected and analyzed for Ph- participants.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Bosutinib: Chronic Phase 2nd Line Chronic Myelogenous Leukemia | Bosutinib: Chronic Phase 3rd Line Chronic Myelogenous Leukemia | Bosutinib: Chronic Phase 4th Line Chronic Myelogenous Leukemia | Bosutinib: Accelerated Phase Chronic Myelogenous Leukemia
Number analyzed (Participants) | 43 | 55 | 45 | 4
percentage of participants
  At 3 months | 81.4 [66.6 to 91.6] | 80.0 [67.0 to 89.6] | 55.6 [40.0 to 70.4] | 75.0 [19.4 to 99.4]
  At 6 months | 69.8 [53.9 to 82.8] | 63.6 [49.6 to 76.2] | 62.2 [46.5 to 76.2] | 25.0 [0.6 to 80.6]
  At 12 months | 69.8 [53.9 to 82.8] | 65.5 [51.4 to 77.8] | 48.9 [33.7 to 64.2] | 25.0 [0.6 to 80.6]
  At 18 months | 67.4 [51.5 to 80.9] | 63.6 [49.6 to 76.2] | 42.2 [27.7 to 57.8] | 25.0 [0.6 to 80.6]
  At 24 months | 67.4 [51.5 to 80.9] | 54.5 [40.6 to 68.0] | 44.4 [29.6 to 60.0] | 25.0 [0.6 to 80.6]

8. Secondary Outcome: Percentage of Accelerated Phase Participants With Confirmed Overall Hematological Response (OHR) at Month 3, 6, 9, 12, 18, and 24
Description: as for outcome 5
Time Frame: Months 3, 6, 9, 12, 18, and 24
Population: Evaluable set hematological response: treated participants with a valid baseline hematologic assessment. Data for this outcome measure was not planned to be collected and analyzed for CP2L, CP3L, CP4L and Ph- CML participants.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Bosutinib: Accelerated Phase Chronic Myelogenous Leukemia
Number analyzed (Participants) | 4
percentage of participants
  At 3 months | 75.0 [19.4 to 99.4]
  At 6 months | 50.0 [6.8 to 93.2]
  At 9 months | 75.0 [19.4 to 99.4]
  At 12 months | 75.0 [19.4 to 99.4]
  At 18 months | 25.0 [0.6 to 80.6]
  At 24 months | 0.0 [0.0 to 60.2]

9. Secondary Outcome: Percentage of Participants With Cumulative Confirmed Complete Hematological Response (CHR)
Description: CHR was defined as WBC <10*10^9/L, peripheral blood basophils <5%, no peripheral blood myelocytes, promyelocytes, myeloblasts in the differential, platelet count <450*10^9/L, spleen not palpable. Hematologic responses must be of >=4 weeks duration confirmed by 2 assessments >=4 weeks apart.
Time Frame: Up to 4 years
Population: Evaluable set for hematological response: treated participants with a valid baseline hematologic assessment. Data for this outcome measure was not planned to be collected and analyzed for Ph- participants.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Bosutinib: Chronic Phase 2nd Line Chronic Myelogenous Leukemia | Bosutinib: Chronic Phase 3rd Line Chronic Myelogenous Leukemia | Bosutinib: Chronic Phase 4th Line Chronic Myelogenous Leukemia | Bosutinib: Accelerated Phase Chronic Myelogenous Leukemia
Number analyzed (Participants) | 46 | 61 | 48 | 4
percentage of participants | 91.3 [79.2 to 97.6] | 82.0 [70.0 to 90.6] | 77.1 [62.7 to 88.0] | 75.0 [19.4 to 99.4]

10. Secondary Outcome: Percentage of Participants With Cumulative Major Molecular Response (MMR)
Description: Molecular response: MR4.5/MR4/MMR defined as <=0.0032/0.01/0.1% BCR-ABL1 ratio respectively, on IS corresponding to >=4.5/4/3-log reduction from standardized baseline with at least 32,000/10,000/10,000 ABL1 assessed by central laboratory. To be considered a responder, the participant must have had maintenance of baseline response while on-treatment or an improvement from baseline.
Time Frame: Up to 4 years
Population: Evaluable set for molecular response: treated participants with a valid baseline molecular assessment. Data for this outcome measure was not planned to be collected and analyzed for Ph- participants.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Bosutinib: Chronic Phase 2nd Line Chronic Myelogenous Leukemia | Bosutinib: Chronic Phase 3rd Line Chronic Myelogenous Leukemia | Bosutinib: Chronic Phase 4th Line Chronic Myelogenous Leukemia | Bosutinib: Accelerated Phase Chronic Myelogenous Leukemia
Number analyzed (Participants) | 46 | 55 | 48 | 4
percentage of participants
  MMR | 82.6 [68.6 to 92.2] | 76.4 [63.0 to 86.8] | 56.3 [41.2 to 70.5] | 50.0 [6.8 to 93.2]
  MR4 | 73.9 [58.9 to 85.7] | 63.6 [49.6 to 76.2] | 41.7 [27.6 to 56.8] | 25.0 [0.6 to 80.6]
  MR4.5 | 58.7 [43.2 to 73.0] | 50.9 [37.1 to 64.6] | 35.4 [22.2 to 50.5] | 25.0 [0.6 to 80.6]

11. Secondary Outcome: Kaplan-Meier Estimate of Probability of Retaining Complete Cytogenetic Response (CCyR) at Month 36
Description: Kaplan-Meier analysis. Duration of CCyR: from first date of CCyR to date of confirmed loss of CCyR/disease progression/on-treatment death or censoring, analyzed for responders only. CyR: prevalence of Ph+ cells. CCyR: 0% Ph+ cells from >=20 metaphases from conventional cytogenetics or <1% Ph+ cells from >=200 cells analyzed by FISH or MMR (<=0.1% BCR-ABL1 on the IS with at least 10,000 ABL1 transcripts assessed by central laboratory). Confirmed loss: 2 consecutive non-response assessments >=28 days apart. Progression: for CP: participants evolving from CP to AP, loss of CHR; loss of MCyR; in participants without CHR WBC >20*10^9/L on 2 occasions >=2 weeks apart after the first 4 weeks of treatment; for AP: confirmed BP, loss of previous hematologic response over a 2-week period, loss of CHR, no decrease from baseline levels (if considered clinically relevant) in percentage blasts in peripheral blood or bone marrow on all assessments over a 4-week period.
Time Frame: At Month 36
Population: Evaluable set for cytogenetic response: treated participants with valid baseline cytogenetic assessment (>= 20 metaphases from baseline bone marrow or CCyR with >=200 cells from FISH or baseline MMR) and who achieved CCyR. Here, "Overall Number of Participants Analyzed" signifies participants evaluable for this outcome measure who had CCyR.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Bosutinib: Chronic Phase 2nd Line Chronic Myelogenous Leukemia | Bosutinib: Chronic Phase 3rd Line Chronic Myelogenous Leukemia | Bosutinib: Chronic Phase 4th Line Chronic Myelogenous Leukemia | Bosutinib: Accelerated Phase Chronic Myelogenous Leukemia
Number analyzed (Participants) | 37 | 46 | 33 | 3
percentage of participants | 96.4 [77.2 to 99.5] | 94.4 [79.2 to 98.6] | 100.0 [100.0 to 100.0] | 100.0 [100.0 to 100.0]

12. Secondary Outcome: Kaplan-Meier Estimate of Probability of Retaining Major Molecular Response (MMR) at Month 36
Description: Kaplan-Meier analysis. Duration of MMR: from first date of MMR to confirmed loss of MMR/disease progression/on-treatment death or censoring, analyzed for responders only. MMR:<=0.1% BCR-ABL1 on the IS with at least 10,000 ABL1 transcripts assessed by central laboratory . Confirmed loss: 2 consecutive non-response assessments >=28 days apart with a <3-log (>0.1%) reduction in transcripts one of which corresponds to a <=2-log reduction (>=1%). Progression: for CP: participants evolving from CP to AP, loss of CHR; loss of MCyR; in participants without CHR WBC >20*10^9/L on 2 occasions >=2weeks apart after the first 4 weeks of treatment; for AP: confirmed BP, loss of previous hematologic response over a 2-week period, loss of CHR, no decrease from baseline levels (if considered clinically relevant) in percentage blasts in peripheral blood or bone marrow on all assessments over a 4-week period.
Time Frame: At Month 36
Population: Evaluable set for molecular response: treated participants with valid baseline molecular assessment and who achieved MMR. Here, "Overall Number of Participants Analyzed" signifies participants evaluable for this outcome measure who had MMR.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Bosutinib: Chronic Phase 2nd Line Chronic Myelogenous Leukemia | Bosutinib: Chronic Phase 3rd Line Chronic Myelogenous Leukemia | Bosutinib: Chronic Phase 4th Line Chronic Myelogenous Leukemia | Bosutinib: Accelerated Phase Chronic Myelogenous Leukemia
Number analyzed (Participants) | 38 | 42 | 27 | 2
percentage of participants | 90.7 [73.9 to 96.9] | 81.5 [63.2 to 91.3] | 90.2 [65.9 to 97.5] | 100.0 [100.0 to 100.0]

13. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs) and Serious AEs
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. TEAE: any event increasing in severity from baseline or any new event started during bosutinib therapy or within 28 days of the last dose of study drug. SAE: an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial/prolonged inpatient hospitalization; life-threatening experience (immediate risk of death); persistent or significant disability/incapacity; congenital anomaly.
Time Frame: First dose of study drug up to 28 days after last dose (up to maximum of 4 years)
Population: The safety analysis set included participants who received at least 1 dose of bosutinib.
Measure: Count of Participants; unit: Participants
Groups:
- Bosutinib: Chronic Myelogenous Leukemia: Participants with Philadelphia chromosome positive chronic phase 2nd, 3rd and 4th line chronic myelogenous leukemia, Philadelphia chromosome positive accelerated phase chronic myelogenous leukemia and BCR-ABL1-chronic myelogenous leukemia/Philadelphia chromosome negative chronic myelogenous leukemia.
Arm/Group | Bosutinib: Chronic Phase 2nd Line Chronic Myelogenous Leukemia | Bosutinib: Chronic Phase 3rd Line Chronic Myelogenous Leukemia | Bosutinib: Chronic Phase 4th Line Chronic Myelogenous Leukemia | Bosutinib: Accelerated Phase Chronic Myelogenous Leukemia | Bosutinib: Philadelphia Chromosome Negative Chronic Myelogenous Leukemia | Bosutinib: Chronic Myelogenous Leukemia
Number analyzed (Participants) | 46 | 61 | 49 | 4 | 3 | 163
Participants
  TEAEs | 46 | 61 | 48 | 4 | 3 | 162
  Treatment-emergent SAEs | 21 | 30 | 14 | 1 | 3 | 69

14. Secondary Outcome: Number of Participants With Grade 3 or 4 Treatment Emergent Adverse Events (TEAEs) Based on National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) Version 4.0
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. TEAE was any event increasing in severity from baseline or any new event that started during bosutinib therapy or within 28 days of the last dose of study drug. Severity was graded as Grade 1: asymptomatic or mild symptoms, clinical or diagnostic observations only, intervention not indicated; Grade 2: moderate, minimal, local or noninvasive intervention indicated, limiting age-appropriate instrumental activities of daily life (ADL); Grade 3: severe or medically significant but not immediately life-threatening, hospitalization or prolongation of existing hospitalization indicated, disabling, limiting self-care ADL; Grade 4: life-threatening consequence, urgent intervention indicated; Grade 5: death related to AE. Number of participants with Grade 3 or 4 TEAEs are reported.
Time Frame: First dose of study drug up to 28 days after last dose (up to maximum of 4 years)
Population: The safety analysis set included participants who received at least 1 dose of bosutinib.
Measure: Count of Participants; unit: Participants
Arm/Group | Bosutinib: Chronic Phase 2nd Line Chronic Myelogenous Leukemia | Bosutinib: Chronic Phase 3rd Line Chronic Myelogenous Leukemia | Bosutinib: Chronic Phase 4th Line Chronic Myelogenous Leukemia | Bosutinib: Accelerated Phase Chronic Myelogenous Leukemia | Bosutinib: Philadelphia Chromosome Negative Chronic Myelogenous Leukemia | Bosutinib: Chronic Myelogenous Leukemia
Number analyzed (Participants) | 46 | 61 | 49 | 4 | 3 | 163
Participants | 36 | 49 | 39 | 2 | 3 | 129

15. Secondary Outcome: Number of Participants With Treatment Related Treatment Emergent Adverse Events (TEAEs)
Description: An AE was any untoward medical occurrence attributed to study drug in a participant who received study drug. TEAE was any event increasing in severity from baseline or any new event that started during bosutinib therapy or within 28 days of the last dose of study drug. Relatedness to drug was assessed by investigator.
Time Frame: First dose of study drug up to 28 days after last dose (up to maximum of 4 years)
Population: The safety analysis set included participants who received at least 1 dose of bosutinib.
Measure: Count of Participants; unit: Participants
Arm/Group | Bosutinib: Chronic Phase 2nd Line Chronic Myelogenous Leukemia | Bosutinib: Chronic Phase 3rd Line Chronic Myelogenous Leukemia | Bosutinib: Chronic Phase 4th Line Chronic Myelogenous Leukemia | Bosutinib: Accelerated Phase Chronic Myelogenous Leukemia | Bosutinib: Philadelphia Chromosome Negative Chronic Myelogenous Leukemia | Bosutinib: Chronic Myelogenous Leukemia
Number analyzed (Participants) | 46 | 61 | 49 | 4 | 3 | 163
Participants | 46 | 61 | 48 | 4 | 3 | 162

16. Secondary Outcome: Number of Participants With Laboratory Abnormalities Based on National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) Version 4.03
Description: Number of participants with any hematological, chemistry and coagulation abnormality of any grade were reported. Hematological: absolute neutrophil count (low), hemoglobin (low), lymphocytes (low), platelets (low) and leukocytes (low). Chemistry: alkaline phosphatase (high), alanine aminotransferase (high), amylase (high), aspartate aminotransferase (high), bilirubin (high), creatinine (high), lipase (high). Coagulation: activated partial prothrombin time (low), prothrombin time (low and high), partial prothrombin time (high).
Time Frame: First dose of study drug up to 28 days after last dose (up to maximum of 4 years)
Population: The safety analysis set included participants who received at least 1 dose of bosutinib.
Measure: Count of Participants; unit: Participants
Arm/Group | Bosutinib: Chronic Phase 2nd Line Chronic Myelogenous Leukemia | Bosutinib: Chronic Phase 3rd Line Chronic Myelogenous Leukemia | Bosutinib: Chronic Phase 4th Line Chronic Myelogenous Leukemia | Bosutinib: Accelerated Phase Chronic Myelogenous Leukemia | Bosutinib: Philadelphia Chromosome Negative Chronic Myelogenous Leukemia | Bosutinib: Chronic Myelogenous Leukemia
Number analyzed (Participants) | 46 | 61 | 49 | 4 | 3 | 163
Participants
  Hematology | 38 | 56 | 40 | 4 | 3 | 141
  Chemistry | 46 | 61 | 49 | 4 | 3 | 163
  Coagulation | 18 | 25 | 12 | 2 | 1 | 58

ADVERSE EVENTS:
Time Frame: From first dose of study drug up to 28 days after last dose (up to maximum of 4 years)
Description: The total number of deaths occurring during study, from first dose and up to the end of the study are reported for all treated participants and includes deaths which occurred after 28 days post last study drug dose. Same event may appear as both an AE and Serious Adverse Events. An event may be categorized as serious in 1 participant and as non-serious in another, or a participant may have experienced both a serious and non-serious event. Analysis performed on safety set.
Arm/Group | Bosutinib: Chronic Phase 2nd Line Chronic Myelogenous Leukemia | Bosutinib: Chronic Phase 3rd Line Chronic Myelogenous Leukemia | Bosutinib: Chronic Phase 4th Line Chronic Myelogenous Leukemia | Bosutinib: Accelerated Phase Chronic Myelogenous Leukemia | Bosutinib: Philadelphia Chromosome Negative Chronic Myelogenous Leukemia | Bosutinib: Chronic Myelogenous Leukemia
All-Cause Mortality (participants affected / at risk) | 5/46 | 7/61 | 5/49 | 0/4 | 2/3 | 19/163
Serious Adverse Events (participants affected / at risk) | 21/46 | 30/61 | 14/49 | 1/4 | 3/3 | 69/163
Other Adverse Events (participants affected / at risk) | 46/46 | 61/61 | 48/49 | 4/4 | 3/3 | 162/163
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bosutinib: Chronic Phase 2nd Line Chronic Myelogenous Leukemia (N=46) | Bosutinib: Chronic Phase 3rd Line Chronic Myelogenous Leukemia (N=61) | Bosutinib: Chronic Phase 4th Line Chronic Myelogenous Leukemia (N=49) | Bosutinib: Accelerated Phase Chronic Myelogenous Leukemia (N=4) | Bosutinib: Philadelphia Chromosome Negative Chronic Myelogenous Leukemia (N=3) | Bosutinib: Chronic Myelogenous Leukemia (N=163)
Anaemia (Blood and lymphatic system disorders) | 1 | 2 | 0 | 0 | 0 | 3
Abdominal lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 1
Pancytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 1
Cardiac failure (Cardiac disorders) | 2 | 3 | 1 | 0 | 0 | 6
Atrial fibrillation (Cardiac disorders) | 3 | 1 | 1 | 0 | 0 | 5
Pericardial effusion (Cardiac disorders) | 2 | 0 | 1 | 0 | 1 | 4
Angina pectoris (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 1
Angina unstable (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 1
Atrioventricular block complete (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 1
Bundle branch block right (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 1
Cardiogenic shock (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 1
Cardiomyopathy (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 1
Coronary artery occlusion (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 1
Sinus node dysfunction (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 1
Keratoconus (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0 | 2
Appendiceal mucocoele (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 1
Ascites (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 1
Colitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 1
Hiatus hernia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 1
Ileus (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 1
Oesophageal fistula (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 1
Rectal polyp (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 1
Subileus (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 1
Pyrexia (General disorders) | 1 | 3 | 0 | 0 | 0 | 4
Chest pain (General disorders) | 0 | 1 | 0 | 0 | 0 | 1
Multiple organ dysfunction syndrome (General disorders) | 1 | 0 | 0 | 0 | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0 | 1
Hepatic cirrhosis (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 1
Hypersensitivity (Immune system disorders) | 0 | 0 | 1 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 2 | 3 | 0 | 0 | 5
Cellulitis (Infections and infestations) | 0 | 0 | 1 | 1 | 0 | 2
Appendicitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 1
Bronchitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 1
Pneumonia pneumococcal (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 1
Pseudomembranous colitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 1
Sepsis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 1
Viral infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 1
Arterial restenosis (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 1
Femur fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 1
Spinal fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 1
Tendon rupture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 1
Blood creatinine increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 1
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 1
Fluid retention (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 1
Metabolic disorder (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0 | 0 | 0 | 3
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 1
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 1
Anaplastic large-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 1
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 1
Laryngeal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 1
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 1
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 1
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 1
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 1
Syncope (Nervous system disorders) | 1 | 1 | 1 | 0 | 0 | 3
Cerebrovascular accident (Nervous system disorders) | 0 | 2 | 0 | 0 | 0 | 2
Transient ischaemic attack (Nervous system disorders) | 1 | 1 | 0 | 0 | 0 | 2
Sciatica (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 2 | 1 | 1 | 0 | 0 | 4
Chronic kidney disease (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 1
Breast mass (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 1
Ovarian cyst ruptured (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 3 | 0 | 1 | 7
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0 | 0 | 0 | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 0 | 2
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 1
Emphysema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 1
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 1
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 1
Peripheral arterial occlusive disease (Vascular disorders) | 0 | 2 | 1 | 0 | 0 | 3
Peripheral ischaemia (Vascular disorders) | 0 | 2 | 0 | 0 | 0 | 2
Haemorrhage (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 1
Shock haemorrhagic (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Bosutinib: Chronic Phase 2nd Line Chronic Myelogenous Leukemia (N=46) | Bosutinib: Chronic Phase 3rd Line Chronic Myelogenous Leukemia (N=61) | Bosutinib: Chronic Phase 4th Line Chronic Myelogenous Leukemia (N=49) | Bosutinib: Accelerated Phase Chronic Myelogenous Leukemia (N=4) | Bosutinib: Philadelphia Chromosome Negative Chronic Myelogenous Leukemia (N=3) | Bosutinib: Chronic Myelogenous Leukemia (N=163)
Anaemia (Blood and lymphatic system disorders) | 7 | 14 | 5 | 0 | 2 | 28
Thrombocytopenia (Blood and lymphatic system disorders) | 7 | 6 | 4 | 1 | 1 | 19
Neutropenia (Blood and lymphatic system disorders) | 3 | 4 | 0 | 0 | 0 | 7
Atrial fibrillation (Cardiac disorders) | 4 | 2 | 0 | 0 | 0 | 6
Cardiac failure (Cardiac disorders) | 3 | 2 | 1 | 0 | 0 | 6
Dry eye (Eye disorders) | 3 | 1 | 1 | 0 | 0 | 5
Conjunctival hyperaemia (Eye disorders) | 3 | 2 | 0 | 0 | 0 | 5
Diarrhoea (Gastrointestinal disorders) | 43 | 54 | 42 | 4 | 2 | 145
Nausea (Gastrointestinal disorders) | 15 | 29 | 25 | 1 | 0 | 70
Vomiting (Gastrointestinal disorders) | 13 | 22 | 19 | 0 | 1 | 55
Abdominal pain (Gastrointestinal disorders) | 14 | 17 | 16 | 2 | 0 | 49
Abdominal pain upper (Gastrointestinal disorders) | 19 | 8 | 9 | 0 | 1 | 37
Constipation (Gastrointestinal disorders) | 13 | 11 | 7 | 0 | 1 | 32
Dyspepsia (Gastrointestinal disorders) | 4 | 6 | 3 | 1 | 0 | 14
Abdominal distension (Gastrointestinal disorders) | 3 | 5 | 3 | 0 | 0 | 11
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 4 | 3 | 2 | 1 | 0 | 10
Flatulence (Gastrointestinal disorders) | 5 | 3 | 1 | 0 | 0 | 9
Abdominal discomfort (Gastrointestinal disorders) | 3 | 2 | 1 | 0 | 0 | 6
Fatigue (General disorders) | 10 | 15 | 19 | 1 | 1 | 46
Asthenia (General disorders) | 20 | 9 | 6 | 1 | 0 | 36
Pyrexia (General disorders) | 7 | 11 | 13 | 0 | 0 | 31
Oedema peripheral (General disorders) | 9 | 11 | 9 | 0 | 0 | 29
Chest pain (General disorders) | 4 | 1 | 0 | 0 | 1 | 6
Influenza like illness (General disorders) | 4 | 1 | 1 | 0 | 0 | 6
Nasopharyngitis (Infections and infestations) | 7 | 11 | 8 | 0 | 0 | 26
Influenza (Infections and infestations) | 6 | 3 | 5 | 0 | 0 | 14
Urinary tract infection (Infections and infestations) | 1 | 6 | 2 | 0 | 0 | 9
Bronchitis (Infections and infestations) | 3 | 3 | 2 | 0 | 0 | 8
Upper respiratory tract infection (Infections and infestations) | 1 | 5 | 2 | 0 | 0 | 8
Folliculitis (Infections and infestations) | 6 | 1 | 0 | 0 | 0 | 7
Fall (Injury, poisoning and procedural complications) | 2 | 10 | 3 | 0 | 0 | 15
Alanine aminotransferase increased (Investigations) | 10 | 18 | 16 | 0 | 0 | 44
Aspartate aminotransferase increased (Investigations) | 9 | 11 | 13 | 0 | 0 | 33
Blood creatinine increased (Investigations) | 8 | 7 | 10 | 1 | 0 | 26
Lipase increased (Investigations) | 9 | 11 | 5 | 0 | 0 | 25
Amylase increased (Investigations) | 5 | 8 | 3 | 0 | 0 | 16
Weight decreased (Investigations) | 2 | 7 | 4 | 0 | 1 | 14
Gamma-glutamyl transferase increased (Investigations) | 3 | 6 | 3 | 0 | 1 | 13
Blood uric acid increased (Investigations) | 1 | 6 | 2 | 0 | 0 | 9
Blood folate decreased (Investigations) | 3 | 2 | 0 | 0 | 0 | 5
Decreased appetite (Metabolism and nutrition disorders) | 4 | 10 | 7 | 1 | 1 | 23
Hyperuricaemia (Metabolism and nutrition disorders) | 3 | 0 | 2 | 0 | 0 | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 8 | 18 | 10 | 0 | 1 | 37
Myalgia (Musculoskeletal and connective tissue disorders) | 7 | 12 | 4 | 0 | 0 | 23
Pain in extremity (Musculoskeletal and connective tissue disorders) | 8 | 8 | 5 | 0 | 1 | 22
Bone pain (Musculoskeletal and connective tissue disorders) | 5 | 4 | 3 | 0 | 1 | 13
Neck pain (Musculoskeletal and connective tissue disorders) | 4 | 4 | 2 | 0 | 0 | 10
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 3 | 1 | 1 | 0 | 0 | 5
Headache (Nervous system disorders) | 14 | 17 | 14 | 2 | 0 | 47
Paraesthesia (Nervous system disorders) | 3 | 1 | 0 | 0 | 1 | 5
Insomnia (Psychiatric disorders) | 4 | 2 | 4 | 0 | 1 | 11
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 9 | 17 | 12 | 0 | 1 | 39
Cough (Respiratory, thoracic and mediastinal disorders) | 8 | 18 | 3 | 1 | 1 | 31
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 6 | 13 | 9 | 0 | 1 | 29
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 10 | 1 | 0 | 0 | 0 | 11
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 4 | 1 | 0 | 0 | 5
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 0 | 0 | 0 | 4
Pruritus (Skin and subcutaneous tissue disorders) | 5 | 6 | 7 | 0 | 0 | 18
Alopecia (Skin and subcutaneous tissue disorders) | 5 | 5 | 2 | 0 | 1 | 13
Dry skin (Skin and subcutaneous tissue disorders) | 3 | 3 | 5 | 2 | 0 | 13
Skin lesion (Skin and subcutaneous tissue disorders) | 4 | 3 | 2 | 0 | 0 | 9
Erythema (Skin and subcutaneous tissue disorders) | 5 | 2 | 1 | 0 | 0 | 8
Acne (Skin and subcutaneous tissue disorders) | 3 | 3 | 1 | 0 | 0 | 7
Rash pruritic (Skin and subcutaneous tissue disorders) | 4 | 3 | 0 | 0 | 0 | 7
Night sweats (Skin and subcutaneous tissue disorders) | 3 | 0 | 1 | 0 | 0 | 4
Hypertension (Vascular disorders) | 4 | 1 | 8 | 1 | 1 | 15
Haematoma (Vascular disorders) | 0 | 4 | 1 | 0 | 0 | 5
Back pain (Musculoskeletal and connective tissue disorders) | 7 | 13 | 9 | 0 | 0 | 29
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 | 5 | 2 | 0 | 2 | 11
Dizziness (Nervous system disorders) | 8 | 9 | 9 | 0 | 1 | 27
Rash (Skin and subcutaneous tissue disorders) | 9 | 8 | 8 | 0 | 0 | 25
Gastrointestinal disorder (Gastrointestinal disorders) | 3 | 1 | 0 | 0 | 0 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2017-09-07): https://cdn.clinicaltrials.gov/large-docs/82/NCT02228382/Prot_000.pdf
  • Statistical Analysis Plan (2020-11-12): https://cdn.clinicaltrials.gov/large-docs/82/NCT02228382/SAP_001.pdf